CLINICAL TRIAL: NCT02631239
Title: The Efficacy and Safety of Etoposide, Dexamethasone, Peg-asparaginase or Plus Methotrexate With Sandwiched Radiotherapy in the Treatment of Stage I to II Extranodal Natural Killer/T-Cell Lymphoma, Nasal Type
Brief Title: MESA Versus ESA in the Treatment of Early Stage NK/T-cell Lymphoma
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Zhao Weili, Professor, Ruijin Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RJ-NK-2015
Record Dates: First submitted 2015-11-28; First posted 2015-12-16 (Estimated); Last update posted 2021-08-25 (Actual); Status verified 2021-08

CONDITIONS: Extranodal NK/T-cell Lymphoma, Nasal Type
MeSH Terms: conditions — Lymphoma, Extranodal NK-T-Cell | interventions — Methotrexate; Etoposide; Dexamethasone; pegaspargase; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- MESA (Active Comparator): Methotrexate, etoposide, dexamethasone, Peg-asparaginase and sandwiched radiotherapy
  Interventions: Drug: Methotrexate; Drug: Etoposide; Drug: Dexamethasone; Drug: Pegaspargase; Radiation: Radiotherapy
- ESA (Experimental): Etoposide, dexamethasone, Peg-asparaginase and sandwiched radiotherapy
  Interventions: Drug: Etoposide; Drug: Dexamethasone; Drug: Pegaspargase; Radiation: Radiotherapy

INTERVENTIONS:
Drug: Methotrexate — 1g/m2/d IV *1d
  Arms: MESA
Drug: Etoposide — 200mg/d PO *3d
Drug: Dexamethasone — 40mg/d PO *3d
Drug: Pegaspargase — 2500IU/m2/d IM *1d
Radiation: Radiotherapy — 50-56Gy

SUMMARY:
Extranodal natural killer (NK)/T-cell lymphoma (ENKTL), nasal type, is a distinct and heterogeneous histopathologic subtype of non-Hodgkin lymphoma (NHL), accounting for 5%~10%. The frequency of ENKTL among NHL patients is significantly higher in Asia than in Western countries, with poor prognosis. Radiotherapy plus chemotherapy has improved the survival for these patients. But the optimal treatment schedule is controversial. The previous protocols usually contained high dose methotrexate, but the application of them is limited for the toxicity.

DETAILED DESCRIPTION:
In mid-2016, we had the final evaluation of the phase 2 study of MESA with sandwiched radiotherapy in newly diagnosed early stage NKTCL (NCT02825147). We obtained the final overall response rate of MESA with sandwiched radiotherapy, while the 2-year progression free survival rate was not available at that timepoint. To make the study design of sample size more accurate, we changed the primary outcome endpoint from 2-year progression free survival rate to overall response rate. The change had been approved by the Ethics Committee in August 10, 2016. At that time, only fourteen patients were enrolled in NCT02631239.

ELIGIBILITY:
Inclusion Criteria:

* Pathological diagnosis of extranodal NK/T cell lymphoma, nasal type, previously untreated
* Age 14 ~ 70 years old
* ECOG(Eastern Cooperative Oncology Group）performance status 0~2
* Stage I to II
* Life expectancy>6 months
* Informed consented

Exclusion Criteria:

* Chemotherapy before
* Bone marrow transplantation before
* History of malignancy
* Uncontrollable cardio-cerebral vascular, coagulative, autoimmune, serious infectious disease
* LVEF≤50%
* Other uncontrollable medical condition that may that may interfere the participation of the study
* Lab at enrollment ALT or AST >3*ULN, AKP or bilirubin >2.5*ULN Creatinine>1.5*ULN
* Not able to comply to the protocol for mental or other unknown reasons
* Pregnant or lactation
* HIV infection

Ages: 14 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 256 (Estimated)
Dates: Start 2016-03-16 (Actual); Primary Completion 2021-03-05 (Actual); Study Completion 2022-07-17 (Estimated)

PRIMARY OUTCOMES:
Overall response rate | 21 days after 4 cycles of chemotherapy

SECONDARY OUTCOMES:
Overall survival | 2-year
Number of Participants With Treatment-Related Adverse Events as Assessed by CTCAE v4.0 | Day 1 of each course and then every 3 months for 2 years
Progression free survival | 2-year

CONTACTS AND LOCATIONS:
Overall Officials: Weili Zhao, Prof, Principal Investigator — Ruijin Hospital
Locations (1):
- Ruijin Hospital, Shanghai, Shanghai Municipality, China